CLINICAL TRIAL: NCT00686777
Title: Low Dose Treatment of Ribavirin in Combination With PEG-IFN Alfa-2b in CHC Patients With genotype1 High Viral Load and Low Body Weight
Brief Title: Pegylated Interferon (PEG-IFN) Alfa-2b and Low Dose Ribavirin for the Treatment of Chronic Hepatitis C Patients With Genotype 1 High Viral Load and Low Body Weight (Study P05172)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05172; JPC-06-320-40
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-IFN + Ribavirin (Experimental): Pegylated Interferon alfa-2b was administered to participants at 1.5 μg/kg subcutaneously once weekly for 48 weeks. Ribavirin was administered orally every day after morning and evening meals for 48 weeks at 400 mg/day.
  Interventions: Biological: Pegylated Interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated Interferon alfa-2b — Pegylated Interferon alfa-2b 1.5 ug/kg SC once weekly for 48 weeks
  Other Names: SCH 54031
Drug: Ribavirin — Ribavirin 400 mg/day orally
  Other Names: SCH 18908

SUMMARY:
The objective is to evaluate the efficacy and safety of the combination therapy with subcutaneous (SC) Pegylated Interferon (PEG-IFN) alfa-2b 1.5 ug/kg/week plus low-dose ribavirin administered for 48 weeks in participants with chronic hepatitis C virus (HCV) who are infected with HCV genotype 1 high viral load, and weigh 50 kg or less.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic hepatitis C.
* Minimum 20 years of age
* Willing to use adequate contraception during the course of the study.
* Participants who can be hospitalized for at least 14 days since treatment initiation.
* Positive for HCV genotype 1 (genotype 1a and 1b) with high viral load (HCV-RNA >=100 kIU/mL).
* Participants weighing over 40 kg to 50 kg.
* Hematology results of:

  * hemoglobin levels >=12 g/dL
  * neutrophils >=1,500/mm^3
  * platelets >=100,000/mm^3

Exclusion Criteria:

* Previous ribavirin therapy.
* Previous interferon therapy within 90 days of registration.
* Participants who received treatment with injectable products containing glycyrrhizin/cysteine/glycine (Stronger Neo-Minophagen C, etc.), Shosaikoto, or ursodeoxycholic acid within 30 days before the start of treatment
* Participants who received treatment with an antiviral or anti-tumor drug or who received immunomodulating therapy (including steroids and radiotherapy) within 90 days before the start of treatment [excluding local administration and topical drugs].
* Participants who received other investigational drugs within 180 days before the start of treatment.
* Hepatitis Bs (HBs) antigen-positive
* Antinuclear antibodies >=1:160
* Fasting blood glucose >=110 mg/dL (however, participants with fasting blood glucose of 110 mg/dL to <126 mg/dL can be registered if HbA1c is <6.5%)
* Participants diagnosed with liver cirrhosis in most recent celioscopy or liver biopsy.
* Participants with or who have a history of any of the following: liver failure; hepatic encephalopathy, esophageal varices, or ascites; depression or schizophrenia requiring treatment or suicidal attempt or ideation; epileptic seizures requiring drug treatment; autoimmune disease (such as Hashimoto's disease, Crohn's disease, ulcerative colitis, chronic rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic erythematosus, autoimmune hemolytic anemia, and scleroderma); hepatic cancer
* Participants with any of the following: liver disease such as autoimmune hepatitis, alcoholic liver disease, and drug-induced hepatic impairment; hemophilia; arrhythmia requiring treatment and participants with or who have a history of angina pectoris, cardiac failure, myocardial infarction, or life-threatening arrhythmia; hypertension (systolic BP of 160 mmHg or more and diastolic BP of 100 mmHg or more) not possible to control with drug therapy; chronic pulmonary disease; hemoglobinopathy (thalassemia, sickle cell anemia); malignant tumor or who have a history of malignant tumor within the past 5 years; thyroid function disorder not controlled by drug therapy.
* Participants with organ transplants (excluding cornea and hair transplants).
* Participants with a history of hypersensitivity to interferon preparations, nucleoside analogs, or biological products such as vaccine.
* Participants with a specific response to PEG-IFN alfa-2b in a prick test to be conducted just before the initiation of treatment.
* Participants who are pregnant or nursing (in the case of male Participants : partner is pregnant)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants could be discontinued from study by meeting prespecified AE discontinuance criteria defined in the protocol. Prespecified adverse event discontinuance criteria included neutrophil count <500 /mm3, platelet count <50,000/mm3, and hemoglobin <8.5 g/dL
Groups:
- Pegylated Interferon Alfa-2b (PEG-IFN) + Ribavirin: PEG-IFN was administered to participants at 1.5 μg/kg subcutaneously once weekly for 48 weeks. Ribavirin was administered orally every day after morning and evening meals for 48 weeks at 400 mg/day.
Period: Overall Study
Arm/Group | Pegylated Interferon Alfa-2b (PEG-IFN) + Ribavirin
Started | 75
Completed 24 Weeks of Treatment | 69
Completed 48 Weeks of Treatment | 65
Included in Follow-up (All Treated) | 75
Completed 24 Weeks of Follow-up | 70
Completed | 65 (Of 10 noncompleters, 6 had AEs including 4 meeting protocol prespecified AE discontinuance criteria.)
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 2
Not completed — Discontinuance Criteria (specified AEs) | 4
Not completed — No Visit | 1

BASELINE CHARACTERISTICS:
Groups:
- PEG-IFN + Ribavirin: PEG-IFN was administered to participants at 1.5 μg/kg subcutaneously once weekly for 48 weeks. Ribavirin was administered orally every day after morning and evening meals for 48 weeks at 400 mg/day.
Arm/Group | PEG-IFN + Ribavirin
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.7)
Age, Customized [Number; unit: participants]
  < 65 yrs | 64
  ≥ 65 yrs | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 24 Weeks After the End of Treatment (EOT) or Discontinuation
Description: SVR was defined as a viral response which was sustained at 24 weeks after the end of treatment as measured by Hepatitis C Virus Ribonucleic Acid (HCV-RNA) negativity.
  HCV-RNA negativity was assessed by an reverse transcriptase polymerase chain reaction (RT-PCR) method, where a negative response was defined by a negative qualitative HCV-RNA result.
Time Frame: Measured at 24 weeks after the end of treatment (at the end of follow-up)
Population: All treated Participants
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN + Ribavirin
Number analyzed (Participants) | 75
percentage of participants | 30.7

2. Secondary Outcome: Percentage of Participants With HCV-RNA Negativity at 24 Weeks of Treatment and at EOT
Description: HCV-RNA negativity was assessed by an RT-PCR method, where a negative response was defined by a negative qualitative HCV-RNA result.
Time Frame: Measured at 24 weeks of treatment and at EOT (Treatment week 48)
Population: All treated Participants
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN + Ribavirin
Number analyzed (Participants) | 75
percentage of participants
  At 24 Weeks Treatment | 61.3
  At End of Treatment | 66.7

3. Primary Outcome: Number of Participants Discontinuing Treatment
Description: Prespecified adverse event discontinuance criteria included neutrophil count <500 /mm3, platelet count <50,000/mm3, and hemoglobin <8.5 g/dL.
Time Frame: From time of first treatment to Week 48
Measure: Number; unit: participants
Arm/Group | PEG-IFN + Ribavirin
Number analyzed (Participants) | 75
participants
  Due To Decrease in Neutrophil Count | 3
  Due To Decrease in Neutrophil and Platelet Count | 1
  Due To Apathy | 1
  Due To Pleural Effusion | 1
  Due To Pregnancy of Participant's Partner | 1
  Due To No Visit | 1
  Due To Withdrawal by Subject | 2
  Total Number Discontinued | 10

ADVERSE EVENTS:
Arm/Group | PEG-IFN + Ribavirin
Serious Adverse Events (participants affected / at risk) | 7/75
Other Adverse Events (participants affected / at risk) | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN + Ribavirin (N=75)
MENINGOCELE (Congenital, familial and genetic disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1)
LABYRINTHITIS (Infections and infestations) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 1 (1)
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
THREATENED LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN + Ribavirin (N=75)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
PALPITATIONS (Cardiac disorders) | 4 (6)
TINNITUS (Ear and labyrinth disorders) | 7 (7)
VERTIGO (Ear and labyrinth disorders) | 4 (5)
ABNORMAL SENSATION IN EYE (Eye disorders) | 8 (8)
ASTHENOPIA (Eye disorders) | 8 (10)
DRY EYE (Eye disorders) | 5 (5)
RETINOPATHY (Eye disorders) | 4 (4)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 18 (20)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (18)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 (15)
CHEILITIS (Gastrointestinal disorders) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 16 (17)
DIARRHOEA (Gastrointestinal disorders) | 26 (43)
GASTRITIS (Gastrointestinal disorders) | 6 (6)
NAUSEA (Gastrointestinal disorders) | 44 (57)
STOMATITIS (Gastrointestinal disorders) | 29 (36)
VOMITING (Gastrointestinal disorders) | 15 (21)
CHEST PAIN (General disorders) | 4 (4)
CHILLS (General disorders) | 11 (11)
FATIGUE (General disorders) | 5 (5)
FEELING COLD (General disorders) | 7 (7)
INJECTION SITE ERYTHEMA (General disorders) | 30 (30)
INJECTION SITE PRURITUS (General disorders) | 26 (26)
INJECTION SITE RASH (General disorders) | 11 (12)
MALAISE (General disorders) | 66 (84)
PAIN (General disorders) | 4 (4)
PYREXIA (General disorders) | 73 (98)
THIRST (General disorders) | 10 (11)
CYSTITIS (Infections and infestations) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 35 (51)
PHARYNGITIS (Infections and infestations) | 4 (4)
CONTUSION (Injury, poisoning and procedural complications) | 4 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 22 (22)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 22 (23)
BASOPHIL COUNT INCREASED (Investigations) | 14 (16)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 5 (5)
BLOOD ALBUMIN DECREASED (Investigations) | 4 (5)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 5 (5)
BLOOD PHOSPHORUS DECREASED (Investigations) | 8 (9)
BLOOD POTASSIUM DECREASED (Investigations) | 14 (15)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 8 (10)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 17 (18)
C-REACTIVE PROTEIN INCREASED (Investigations) | 6 (8)
EOSINOPHIL COUNT INCREASED (Investigations) | 20 (28)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 16 (16)
HAEMATOCRIT DECREASED (Investigations) | 58 (62)
HAEMOGLOBIN DECREASED (Investigations) | 58 (65)
LYMPHOCYTE COUNT DECREASED (Investigations) | 71 (83)
LYMPHOCYTE COUNT INCREASED (Investigations) | 21 (24)
MONOCYTE COUNT INCREASED (Investigations) | 4 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 69 (90)
NEUTROPHIL COUNT INCREASED (Investigations) | 8 (14)
PLATELET COUNT DECREASED (Investigations) | 43 (53)
RED BLOOD CELL COUNT DECREASED (Investigations) | 59 (63)
RETICULOCYTE PERCENTAGE DECREASED (Investigations) | 7 (10)
RETICULOCYTE PERCENTAGE INCREASED (Investigations) | 34 (43)
THYROXINE FREE DECREASED (Investigations) | 6 (6)
TRI-IODOTHYRONINE FREE DECREASED (Investigations) | 8 (9)
TRI-IODOTHYRONINE FREE INCREASED (Investigations) | 5 (5)
WEIGHT DECREASED (Investigations) | 34 (35)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 73 (83)
DECREASED APPETITE (Metabolism and nutrition disorders) | 54 (66)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 50 (63)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 (20)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 9 (9)
MYALGIA (Musculoskeletal and connective tissue disorders) | 49 (64)
DIZZINESS (Nervous system disorders) | 17 (23)
DIZZINESS POSTURAL (Nervous system disorders) | 5 (6)
DYSGEUSIA (Nervous system disorders) | 17 (18)
HEADACHE (Nervous system disorders) | 68 (86)
HYPOAESTHESIA (Nervous system disorders) | 5 (7)
INSOMNIA (Psychiatric disorders) | 43 (56)
MOOD ALTERED (Psychiatric disorders) | 4 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (19)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 (19)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 6 (8)
ALOPECIA (Skin and subcutaneous tissue disorders) | 63 (64)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (6)
ECZEMA (Skin and subcutaneous tissue disorders) | 10 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 36 (41)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 12 (12)
RASH (Skin and subcutaneous tissue disorders) | 41 (49)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No